CLINICAL TRIAL: NCT06413160
Title: The Cardiovascular-Renal-Metabolic (CRM) Syndrome Survey in Jordan
Acronym: JoCRMSSurvey
Status: Not yet recruiting | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Collaborators: Cardiovascular Academy (Unknown); The Association of Jordanian Medical Laboratory Specialists AJMLS (Unknown)
Responsible Party: Principal Investigator, Ayman J Hammoudeh, MD, FACC, Director, Department of Clinical Research, Jordan Collaborating Cardiology Group
Other Study IDs: CVA/JoCRM-2/2024
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular-renal-metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Centrifuged plasma obtained from peripheral blood sample of the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular-renal-metabolic (CRM) syndrome is defined as a systemic disorder with a collection of related signs and symptoms attributable to the coexistence of multiple cardiovascular, renal and metabolic disease with a common underlying pathophysiology in one individual. Surveying this syndrome in a large population in Jordan aims at studying the risk factors, components and stages of the syndrome, thus helping early screening, diagnosing and treating disease and its risk factors.

DETAILED DESCRIPTION:
Cardiovascular-renal-metabolic (CRM) syndrome is defined as a systemic disorder with a collection of related signs and symptoms attributable to the coexistence of multiple cardiovascular, renal and metabolic disease with a common underlying pathophysiology in one individual.

CRM syndrome reflects the intersection of cardiovascular disease with chronic kidney disease (CKD), and metabolic disease and risk factors (RF). A critical combination of these diseases and their risk factors in the same individual has a profound impact on quality of life and overall mortality. The clinical implications of the presence of CRM are significant, with premature morbidity and mortality, multiple organ-system disease, and high health care budgets mainly driven by the burden of cardiovascular disease (CVD).

There are high prevalence rates of all components of CRM and its RF on a global level and in the Middle East. Of note is the high prevalence of CV in the young, smoking, diabetes mellitus, obesity and dyslipidemia.

The current study will evaluate the prevalence of components and RF of CRM disease in a large population in North, central and South of Jordan.

In the Middle East, no systematic study has evaluated the definition of CRM, definition of its stages, and prevalence of its RF and its relation to the coexisting social determinants of health.

The study will provide new and contemporary knowledge on the definition, staging, and comprehensive approaches to care for patients with CRM, and subsequently exploring opportunities for prevention and care optimization by life style modification and pharmacotherapy.

There are different aspects that explain the interaction between the components of CRM. (A) The bidirectional association between the heart failure and the kidneys (cardiorenal syndrome) in addition to the risk of CAD in patients with CKD, (B) adipose tissue link to atherosclerosis mediated by inflammation, insulin resistance and endothelial dysfunction, and risk for DM (C) DM link to CVD, heart failure and kidney dysfunction., and many other links as well.

Screening for CRM is an important pillar in promoting health in every community. The CRM staging system facilitates identifying individuals at progressive levels of severity starting from the preclinical phase to delay or avoid the onset of clinical CVD and CKD. To appropriately find individuals at stage 0 (i.e., asymptomatic stage) it is important to undertake active screening within the population.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and above).
* Willing to sign an informed consent.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive individuals (N=10,000) visiting allocated medical laboratories in North, Center, and South sections of the country during public free blood testing campaigns planned in August 2024 to June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiovascular-renal-metabolic syndrome | From date of study entry through study completion, an average of 1 year
  1. CVD A. Coronary heart disease: Silent and clinical CAD (chronic stable coronary disease, acute coronary disease [ST-elevation myocardial infarction and non-ST-elevation acute coronary syndrome].
     B. Heart failure. C. Atrial fibrillation. D. Stroke. E. Peripheral artery disease
  2. Renal: chronic kidney disease
  3. Metabolic:
  A. Obesity/ B. Diabetes mellitus (DM).

SECONDARY OUTCOMES:
Elevated levels of blood markers | From date of study entry through study completion, an average of 1 year
  Elevated level of lipoprotein (a) , homocysteine, high sensitivity C-Reactive Protein, insulin resistance, and Urine Creatinine/Albumin ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hammoudeh, MD, FACC, Study Director — Istisjhari Hospital; Imad A Alhaddad, MD, FACC, Study Chair — Jordan Hospital
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No